CLINICAL TRIAL: NCT03347929
Title: NSAIDs in Sciatica (NIS), an Investigator Initiated Randomised Placebo Controlled Trial of Naproxen
Brief Title: NSAIDs in Sciatica NSAIDS IN SCIATICA
Acronym: NIS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ostfold Hospital Trust (Other)
Collaborators: Vestre Viken Hospital Trust (Other); Sykehuset Telemark (Other Government); Helse Stavanger HF (Other Government); Oslo University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SO-2017-1; 2014-003623-21 (EudraCT Number)
Record Dates: First submitted 2017-10-05; First posted 2017-11-20 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-07

CONDITIONS: Sciatica
MeSH Terms: conditions — Sciatica | interventions — Naproxen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Naproxen (Experimental): Naproxen 500 mg twice daily
  Interventions: Drug: Naproxen 500 Mg
- Placebo (Placebo Comparator): Placebo 1 tablet twice daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Naproxen 500 Mg — 10 days treatment with Naproxen 500 mg twice daily
  Arms: Naproxen
Drug: Placebo — 10 days treatment with Placebo1 tablet twice daily
  Arms: Placebo

SUMMARY:
This study will evaluate whether treatment with Naproxen 500 mg twice daily is superior to placebo for the improvement of leg pain in patients with sciatica. Half of patients will receive Naproxen while the other half will receive placebo.

DETAILED DESCRIPTION:
Sciatica is an established term for pain radiating from the lower back or buttock into the leg, commonly caused by a disc herniation. Given their analgesic and anti-inflammatory mechanisms of action, NSAIDs (Non-steroidal anti-inflammatory drugs) have been, and are still being regarded as standard therapy for sciatica.

However, very few randomised controlled trials of NSAIDs have been undertaken in sciatica, and no study has showed clinically meaningful effects as compared to placebo.

Since NSAIDs involve the risk of serious gastrointestinal, vascular and renal side effects there is a strong need to clarify their potential beneficial effects in sciatica.

ELIGIBILITY:
Inclusion criteria:

* Age ≥ 18 years
* Radiating pain below the knee with a severity score of ≥4 on a 0-10 (NRS) in the previous 24 hours
* Signs of nerve root/spinal nerve involvement as indicated by at least one of the following features; myotomal weakness, dermatomal sensory disturbances (e.g. sensory loss, self-reported tingling/numbness), diminished reflexes, radiating pain exacerbation by SLR

Exclusion criteria:

* Not able to read or speak Norwegian.
* Unlikely to adhere to treatment and/ or complete follow-up (e.g ongoing serious psychiatric disease, drug abuse, plans to move)
* Sciatica of known cause other than disc herniation or degenerative stenosis.
* Neurogenic claudication, i.e. pain in the legs on walking or standing that resolves with sitting down or lumbar flexion.
* Symptoms indicating immediate surgery: cauda equina syndrome or a progressive large paresis.
* Women who attempt to conceive, are pregnant or breastfeeding.
* Previous episodes of asthma, urticaria or allergic-type reactions after taking aspirin or other NSAIDs.
* Active or history of peptic ulceration, gastrointestinal bleeding, or perforation.
* Use of drugs known to increase upper gastrointestinal adverse events in combination with Naproxen: anticoagulants, aspirin (acetyl salicylic acid), serotonin reuptake inhibitors and systemic corticosteroids.
* Hepatic enzyme (ASAT/ALAT) values above 1,5 x upper limit of normal (ULN)
* Renal function tests (creatinin/eGFR) outside normal range
* Congestive heart failure, established ischaemic heart disease, peripheral arterial disease, and/or cerebrovascular disease.
* Known hypersensitivity to Naproxen or any of the excipients (lactose, maize starch, povidone, sodium starch glycolate, talcum, magnesium stearate, polysorbate 80)
* Ongoing treatment with aspirin, systemic corticosteroids, diuretics, ACE-inhibitors, lithium and anticoagulants
* Scheduled for spinal surgery prior to end of study
* Reservation against intake of gelatine (the capsules contains gelatine, which among other things is produced by ingredients from pigs)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2017-11-30 (Actual); Primary Completion 2023-06-22 (Actual); Study Completion 2023-06-22 (Actual)

PRIMARY OUTCOMES:
Leg pain | Daily from baseline to day10
  A 0-10 numeric rating scale of average leg pain intensity in the previous 24 hours

SECONDARY OUTCOMES:
Back pain | Daily from baseline to day10
  24 h average back pain will be assessed by a 0-10 numeric rating scale
Disability | Day 0, day 5, day, day 10, day 12
  Roland Morris Disability Questionnaire modified for use in sciatica
Sciatica symptoms | Day 0, day 5, day, day 10, day 12
  Sciatica Bothersomeness Index
Work | Day 0, day 10, day 12
  Ability to work and study as normal
Improvement | Day 5, day 10
  Global perceived change of sciatica/back problem on a verbal rating scale (Completely gone, much better, better, a little better, no change, a little worse, worse and much worse).
Rescue medication | Daily from day1 to day10
  Intake of Paracetamol 500 mg tablets (rescue medication) for pain
Opioid medication | Daily from day1 to day10
  Intake of opioid medication (weak or strong) for pain
Responder | Day 5, day 10
  >30% and >50% reduction in leg pain relative to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Waleed Ghanima, MD,PhD, Study Director — Ostfold Hospital Trust; Anne Haugen, MD,PhD, Principal Investigator — Ostfold Hospital Trust
Locations (4):
- Norway (4):
  - Revmatologisk avdeling, Sykehuset Østfold Moss, Moss
  - Avdeling for fysikalsk medisin og rehabilitering, Oslo University Hospital, Oslo
  - Fysikalsk medisinsk poliklinikk, Sykehuset Telemark, Porsgrunn
  - Avdeling for fysikalsk medisin og rehabilitering, Stavanger Universitetssjukehus, Stavanger

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Grovle L, Hasvik E, Holst R, Saetre A, Brox JI, Mathiassen S, Myhre K, Holmgard TE, Haugen AJ. Efficacy of naproxen in patients with sciatica: multicenter, randomized, double-blind, placebo-controlled trial. Pain. 2024 Nov 1;165(11):2606-2614. doi: 10.1097/j.pain.0000000000003280. Epub 2024 Jun 4. PMID 38833590
- [Derived] Grovle L, Hasvik E, Holst R, Haugen AJ. NSAIDs in sciatica (NIS): study protocol for an investigator-initiated multicentre, randomized placebo-controlled trial of naproxen in patients with sciatica. Trials. 2022 Jun 14;23(1):493. doi: 10.1186/s13063-022-06441-3. PMID 35701830

DOCUMENTS (2):
  • Study Protocol (2022-01-20): https://cdn.clinicaltrials.gov/large-docs/29/NCT03347929/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-15): https://cdn.clinicaltrials.gov/large-docs/29/NCT03347929/SAP_002.pdf